CLINICAL TRIAL: NCT03120273
Title: A Phase 1 Clinical Trial to Evaluate Pharmacokinetics (PK), Pharmacodynamics (PD), and Safety in Healthy Chinese Adults After Multiple Intravenous Administration of Dexlansoprazole
Brief Title: A Clinical Trial to Evaluate the Safety and Tolerability of Dexlansoprazole Injection in Healthy Chinese Adults（Part 2）
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Jiangsu Aosaikang Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASKC263-LC-1-2
Record Dates: First submitted 2017-03-28; First posted 2017-04-19 (Actual); Last update posted 2017-04-19 (Actual); Status verified 2017-03

CONDITIONS: Effect of Drugs; Safety Issues
MeSH Terms: interventions — Dexlansoprazole; Lansoprazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexlansoprazole Injection (Experimental): 15mg q12h,30mg q12h,15mg qd,30mg qd in dexlansoprazole treatment arm for 5 days
  Interventions: Drug: Dexlansoprazole Injection
- Lansoprazole Injection (Active Comparator): 30 mg q12h in lansoprazole treatment arm for 5 days.
  Interventions: Drug: Lansoprazole Injection

INTERVENTIONS:
Drug: Dexlansoprazole Injection — 15mg q12h,30mg q12h,15mg qd,30mg qd for 5 days
  Arms: Dexlansoprazole Injection
Drug: Lansoprazole Injection — 30 mg q12h for 5 days.
  Arms: Lansoprazole Injection

SUMMARY:
This is a single center, open-label, multiple-dose phase 1 clinical trial. This study will determine the pharmacokinetics (PK), pharmacodynamics (PD), safety and side-effect profile of an investigational dexlansoprazole injection after multiple intravenous administration in healthy Chinese adults.

DETAILED DESCRIPTION:
This is a single center, open-label, multiple-dose clinical trial. 5 dosing groups were designed, including 15mg q12h,30mg q12h,15mg qd,30mg qd in dexlansoprazole treatment arm for 5 days, and 30 mg q12h in an active comparator, lansoprazole, treatment arm for 5 days. The study will enroll approximately 70 participants with 14 cases in each group. Participants will make 3 visits to the clinic including 8-day of confinement to the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 Years;
* Male (weight ≥50kg) or female (weight ≥45kg);
* Body mass index (BMI) between 19~28 kg/m2;
* In good health as determined by a physician/investigator based on medical history, vital signs, electrocardiogram (ECG), laboratory tests and physical examination findings at screening;
* Subject who totally understand the aim and progress of this clinical trial, make decision by his/her free will, and signed a consent form to follow the progress;
* Female participant of childbearing potential must have a negative serum pregnancy test at screening, and agrees to use routinely adequate contraception from signing of informed consent throughout the duration of the study and for 6 months following the last dose of study drug;
* Male participant agrees to use adequate contraception and have no plan to donate sperm from signing of informed consent form throughout the duration of the study and for 6 months after the last dose of study drug;
* In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.

Exclusion Criteria:

* Positive breath test result for H pylori at Screening;
* Cannot tolerate placement of the pH probe;
* Has poor peripheral venous access;
* Allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator;
* Subject who has past or present history of any serious diseases, including (but not limited to) digestive, cardiovascular, respiratory, urinary, musculoskeletal, endocrine, psychiatric or neurological, hematologic, immunological or metabolic disorders;
* Human immunodeficiency virus(HIV), hepatitis B virus(HBV), or syphilis positive;
* Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse (defined as alcohol consumption exceeding 14 units per week) within 6 months preceding this study or is unwilling to agree to abstain from alcohol and drugs throughout the study;
* Heavy smokers (>5 cigarettes per day) within 6 months preceding this study or is unwilling to agree to abstain from smoking throughout the study;
* Participation in another study with an investigational drug within the last 3 months preceding this study;
* Blood donation within the last 2 months (>= 400 ml), or have a plan to donate blood within 1 month after this study;
* Intake of any other drug which might influence the results of the trial during two weeks previous to the start of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2017-05-05 (Estimated); Primary Completion 2017-08-31 (Estimated); Study Completion 2017-09-30 (Estimated)

PRIMARY OUTCOMES:
Percentage time with the intragastric potential of hydrogen (pH)>4 | 24 hours post-dose on Day 5
  Duration of intragastric pH>4 within 24 hours postdose
Percentage time with the intragastric pH>6 | 24 hours post-dose on Day 5
  Duration of intragastric pH>6 within 24 hours postdose
The time of the intragastric pH reaching 4 | 12 hours post-dose on Day 5
  The time of intragastric pH reaching 4 after the last dose
The time of the intragastric pH reaching 6 | 12 hours post-dose on Day 5
  The time of intragastric pH reaching 6 after the last dose

SECONDARY OUTCOMES:
Mean intragastric pH | 24 hours post-dose on Day 5
  Mean intragastric pH
Mean intragastric pH per hour | 24 hours post-dose on Day 5
  Mean intragastric pH per hour
Percentage time with the intragastric pH>4 during the first 4 hours | 4 hours post-dose on Day 5
  Duration of intragastric pH>4 within first 4 hours postdose
Percentage time with the intragastric pH>6 during the first 4 hours | 4 hours post-dose on Day 5
  Duration of intragastric pH>6 within first 4 hours postdose
Percentage of the participants with duration time of intragastric pH>4 over 12h | 12 hours post-dose on Day 5
  Numbers of participants with duration time of intragastric pH>4 over 12h
Percentage of the participants with duration time of intragastric pH>6 over 12h | 12 hours post-dose on Day 5
  Numbers of participants with duration time of intragastric pH>6 over 12h
Cmax on day 1 | 12 hours post-dose on Day 5
  Maximum observed plasma concentration for dexlansoprazole
Cmax on day 5 | 12 hours post-dose on Day 5
  Maximum observed plasma concentration for dexlansoprazole
Area under the plasma concentration-time curve (AUC) on day 1 | 12 hours post-dose on Day 5
  AUC from time 0 to the time of the last quantifiable concentration on day 1
AUC(0-12h) on day 5 | 12 hours post-dose on Day 5
  AUC from time 0 to the time of the last quantifiable concentration on day 5
AUC(0-inf) on day 1 | 12 hours post-dose on Day 5
  AUC from time 0 to extrapolated to infinity on day 1
AUC(0-inf) on day 5 | 12 hours post-dose on Day 5
  AUC from time 0 to extrapolated to infinity on day 5

CONTACTS AND LOCATIONS:
Overall Officials: Lihua Wu, Doctor, Principal Investigator — Zhejiang University
Locations (1):
- First affiliated hospital of Zhejiang University, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Wu L, Liu J, Zheng Y, Zhai Y, Lin M, Wu G, Lv D, Shentu J. Pharmacokinetic/Pharmacodynamic Evaluation of Dexlansoprazole Infusion Injection Compared with Lansoprazole in Healthy Chinese Adults. Clin Drug Investig. 2019 Oct;39(10):953-965. doi: 10.1007/s40261-019-00824-2. PMID 31338800